CLINICAL TRIAL: NCT05541354
Title: Simulation for Operating Room Ergonomics - The SORE Study: Creating an Inter-disciplinary Simulation Curriculum for Operating Room Ergonomics
Brief Title: Simulation for Operating Room Ergonomics
Acronym: SORE
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 5471
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Occupational Injuries
Keywords: Ergonomics; Simulation; Medical Education
MeSH Terms: conditions — Occupational Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Stakeholder Interviews: Semi-structured, open-ended interviews will be conducted via Zoom with a purposive sample of surgeons, anesthesiologists and OR nurses and trainees to identify perceived OR ergonomics issues among stakeholders
- OR Observations: Live observation of OR teams by teams of two observers (an anthropologist and an ergonomics expert, such as a chiropractor or physiotherapist). This will be done, in addition to the interview studies, to identify unperceived and misperceived needs using an observation data collection tool. Each of the following 4 phases of surgery will be assessed individually: 1) OR preparation (team arrival to wheels-in), 2) wheels-in to incision, 3) incision to closure, and 4) closure to wheels-out.
- Curriculum Piloting: Participating OR teams will take part in piloting sessions of the developed simulation curriculum to determine if it meets the proposed content objectives and ensure environmental validity.

SUMMARY:
Ergonomics is the study of how people interact with, and work within an environment. This idea is especially important in a setting such as the operating room (OR), which can be both physically and mentally challenging. Poor ergonomic practices lead to physical discomfort and injuries in >50% of OR staff (surgeons, anesthesiologists, and nurses), impacting OR staff quality of life and leading to staff burnout and early retirement. The end result of which is reduced access to care for patients. Furthermore, the added mental effort of dealing with discomfort and pain can also increase the risk of errors and complications, affecting patient outcomes.

Despite high ergonomic stresses in the OR, and the existence of proven recommendations to address them, only a small number of OR staff are aware of ergonomic solutions and how to apply them. To bridge this gap between knowledge and application, we will assess the ergonomic needs of OR teams and develop an educational simulation curriculum to teach ergonomic recommendations to OR teams (surgery, anesthesiology, and nursing staff and trainees).

DETAILED DESCRIPTION:
The Operating Room (OR) is a complex environment with many ergonomic stresses, including those related to patient movement, operative/anesthetic equipment, and surgical bed positioning. Systematic assessments of OR workload have shown that physical demands are at least as high as mental demands for OR teams.

Poor ergonomic management contributes to the high rate of musculoskeletal symptoms (e.g. neck stiffness and back pain) reported by surgeons, OR nurses, and anesthesiologists. These symptoms impact attentional resources and decision-making, increasing the risk of errors and complications. Furthermore, work-related musculoskeletal disorders lead to absenteeism, reduced career longevity, and burnout.

Ergonomic recommendations and interventions for OR staff, including table height adjustments, patient positioning, and placement of equipment, have been developed and proven effective. However, their usefulness is limited by a general lack of awareness and education among OR teams. Despite this, few formalized ergonomic education programs exist.

Furthermore, existing education programs address ergonomics at the individual-level only, and do not consider the interprofessional team environment, potentially limiting effectiveness. Team influence on ergonomics is reliant on non-technical skills such as communication and situational awareness. However, a busy OR environment, where the focus is rightly on patient safety, does not lend itself well to teaching ergonomic principles or providing live feedback. Fortunately, simulation-based training has repeatedly been shown to be an effective teaching tool for such skills. Simulation-based training is also generally positively perceived by medical learners.

With regard to ergonomics specifically, there is emerging evidence that simulation-based teaching can lead to improvements in focused areas of care, such as patient transfer. However, there is currently no simulation curriculum to teach operative ergonomics overall or as a team-based approach. Thus, comprehensive, interprofessional educational programs are needed to increase both awareness and application of ergonomics in the OR. Our study will build an interprofessional, team simulation curriculum involving surgery, anesthesiology, and nursing staff and trainees to address this critical gap in training.

Objectives

1. Assess the perceived and unperceived ergonomic needs of OR teams (surgical, anesthesiology, and nursing staff and trainees).
2. Develop and pilot an interdisciplinary OR ergonomics simulation curriculum for OR teams.

This exploratory study will take part in 2 Phases.

In Phase I, an interprofessional working group with representatives from surgery, anesthesiology, nursing, physiotherapy, chiropractic, medical education, simulation, and human factors engineering will identify gaps in OR ergonomics to inform the creation of the curriculum. Three strategies will be used to identify problems and assess needs in OR ergonomics: 1) initial literature review; 2) semi-structured stakeholder interviews, 3) direct observation of OR teams performing surgical procedures.

Phase II will involve development and piloting of the educational simulation curriculum with OR teams.

ELIGIBILITY:
Inclusion Criteria:

* Member of an OR team (surgery, anesthesiology or nursing staff or trainee) at Sunnybrook Health Sciences Centre

Exclusion Criteria:

* Lack of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A purposive sample of OR stakeholders/teams, including surgeons, anesthesiologists, OR nurses and trainees.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of OR ergonomics simulation curriculum | 18-24 months
  The success of this project will be measured primarily by its development of the final product: an interdisciplinary simulation curriculum for OR ergonomics, with accompanying implementation tools (e.g. website), which is ready to be implemented

SECONDARY OUTCOMES:
Ability to obtain peer reviewed funding for effectiveness study | 18-24 months
  Additional success would be measured by obtaining peer-reviewed funding for a multi-institution implementation and effectiveness assessment of the curriculum.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Research Institute, Toronto, Canada